CLINICAL TRIAL: NCT00755664
Title: Effects of Low-dose B-vitamins Supplementation on Plasma Homocysteine and Framingham Risk Score: Double Blind Randomized Controlled Trial in Healthy Chinese Elderly
Brief Title: Effects of Low-dose Complex B-vitamins on Homocysteine and Framingham Risk Score Among Chinese Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Institute of reproductive and Child Health (Unknown); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Liu Jianmeng, Institute of reproductive and Child Health, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 30572071
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Hyperhomocysteinemia
Keywords: homocysteine; folate acid,; vitamin B; random controlled trail
MeSH Terms: conditions — Hyperhomocysteinemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose complex B-vitamins (Active Comparator): Intervention group receives Low-dose complex B-vitamins every day. Low-dose complex B-vitamins contain 400µg of folic acid, 2mg of vitamin B6, 10µg of vitamin B12 and 50mg vitamin C. Daily supplementation lasts for 12 months
  Interventions: Dietary Supplement: Low-dose complex B-vitamins
- Vitamin C (Placebo Comparator): Control group receives Vitamin C (50mg)every day. Daily supplementation lasts for 12 months.
  Interventions: Dietary Supplement: Low-dose complex B-vitamins

INTERVENTIONS:
Dietary Supplement: Low-dose complex B-vitamins — The complex B vitamins supplement has been made as capsule and packaging 31 capsules in 1 bottle with a pre-determined code number on its cover. The main content contains either vitamin C 50mg alone or combination with folate 0.4 mg, vitamin B6 2mg, vitamin B12 10μg and vitamin C 50 mg. Two kinds of the supplements could not be discriminated by appearance, smell, taste, size and package.volunteers in either arms are required to take 1 capsule per day and last for 48 weeks.
  Other Names: vitamin supplement

SUMMARY:
The purpose of this study is to evaluate whether low dose complex B-vitamins (folic acid,vitamin B6 and vitamin B12) can lower the risk of developing hyperhomocysteinemia in an apparently healthy population with low folate/B12 and high Hcy status.

DETAILED DESCRIPTION:
Hyperhomocysteinemia has been well known as an independent risk factor for CVD. Numerous studies have demonstrated that certain kinds of vitamin B(folic acid,vitamin B6 and vitamin B12)can reduce Hcy level and may prevent CVD. However, the majority of those studies has been conducted always used high dose vitamin in patient or high risk population. There is thus absence of data that the effectiveness of low dose complex B-vitamins on the apparently Chinese elderly population with relative sub-nutritional status. Our study is just focus on the aforementioned aspect.

ELIGIBILITY:
Inclusion Criteria:

* Male and female residents living in the field site for at least 12 months
* Aged 60-74 years

Exclusion Criteria:

* History of chronic disease and taking medications for treatment such as CVD, COPD, cancer, severe renal and liver disease, diabetes.
* Use of multivitamins, and individual vitamins such as folic acid, B12, or B6 in the last 6 months.
* Taking medications known to interfere with folate metabolism, including methotrexate, tamoxifen, L-DOPA, niacin, phenytoin, bile acid sequestrants; anticonvulsant medications (such as dilantin, phenytoin, and primidone), Metformin, Sulfasalazine.
* Conditions that prevent participation or compliance such as Downs syndrome, mental problems, or severe cognitive impairment

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
plasma homocysteine level, plasma folate acid and red blood cell folate acid, Framingham risk score | 6,12 and 18 months

SECONDARY OUTCOMES:
systolic blood pressure, diastolic blood pressure and hemoglobin | 6 and 12 months

OTHER OUTCOMES:
folate receptor antibodies | 6 months
genetic variants | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianmeng Liu, Prof., Principal Investigator — Institute of reproductive and Child health, PUHSC
Locations (1):
- The maternal and Children health care hospital, Yuanshi County of Shijiazhuang, Hebei, China